CLINICAL TRIAL: NCT07238335
Title: Comparative Study Between Digital Pick-up of Attachments Before Registration of Jaws Relations and Intraoral Pick-up With Digitally Constructed 2-Implant Mandibular Overdenture Bases : Peri-Implant Alveolar Bone Height Changes
Brief Title: Comparison Between Digital And Direct Pickup Of Attachments With Digitally Constructed 2-Implant Overdenture Bases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nesma mousa, master degree, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A05010023RP
Record Dates: First submitted 2025-09-23; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Estimation of Bone Height Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital pickup before jaw relation (Experimental)
  Interventions: Device: digital pickup of attachment before jaw relation
- intraoral pickup during insertion (Active Comparator)
  Interventions: Device: intraoral pickup of attachment during insertion

INTERVENTIONS:
Device: digital pickup of attachment before jaw relation — Arm 1 - Digital Pick-up Before Jaw Relation
  Intervention Type: Device Description (short): Extraoral digital pick-up of ball attachments on master cast, CAD/CAM denture base fabrication, jaw relation registration, and denture insertion.
  Arms: digital pickup before jaw relation
Device: intraoral pickup of attachment during insertion — Arm 2 - Intraoral Pick-up During Insertion
  Intervention Type: Device Description (short): Intraoral direct pick-up of ball attachments during denture insertion after CAD/CAM denture base fabrication and jaw relation registration.
  Arms: intraoral pickup during insertion

SUMMARY:
Comparing digital attachment pickup prior to jaw relation registration with intraoral pickup using digitally constructed mandibular overdenture bases is the aim of this study.

ELIGIBILITY:
Inclusion Criteria:

* Upper and lower ridges covered with healthy mucosa
* Sufficient quality and quantity of alveolar bone
* Sufficient inter arch space
* Angle class one relation

Exclusion Criteria:

* Active cancer
* Immune disease
* Uncontrolled diabetes

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Peri-implant marginal alveolar bone height using digital periapical radiograph at baseline (definite insertion), 6 months, ,and 12 months after insertion | at baseline (definite insertion), at 6 months, and after 12 months after insertion

CONTACTS AND LOCATIONS:
Overall Officials: mohamed m foaud, phd, Principal Investigator — faculty of dentistry Mansoura university removable Prosthodontics department
Locations (1):
- Faculty of Dentistry Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided